CLINICAL TRIAL: NCT05693662
Title: The Effect of Mindfulness-Based Self-Compassion Education Given to Parents of Children With Autism Spectrum Disorder on Stress, Psychological Resilience and Well-Being
Brief Title: The Effect of Mindfulness-Based Self-Compassion Education Given to Parents of Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mine CENGİZ, Lecturer, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MCENGİZ
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Autism Spectrum Disorder
Keywords: Awareness, well-being, self-compassion, resilience, stress
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: For randomization, parents were randomly assigned to experiment and control by using a computer program module used in randomized controlled studies (https://www.random.org/). Parents of children with ASD are numbered in the order in which they arrived at the hospital. This process was carried out until the experimental and control groups were completed. Parents of children with ASD included in the study were randomized using a single-blind randomization rule. Parents who met the sampling criteria for randomization were ranked up to 68.
Who Masked: Participant, Outcomes Assessor
Masking Description: It was not stated to the parents whether they were in the experimental or control group. It was performed in a single blind manner.The statistician is also blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Session 1 (Experimental): Educational About Autism Spectrum Disorder
  Interventions: Behavioral: Session 1
- Session 2 (Experimental): Mindfulness Based Self-Compassion information
  Interventions: Behavioral: Session 2
- Session 3 (Experimental): How We Evolved - Threat, Impulse, and Soothing Systems
  Interventions: Behavioral: Session 3
- Session 4 (Experimental): Threat and Self-Compassion
  Interventions: Behavioral: Session 4
- Session 5 (Experimental): Untying the Knots of Desires and Patterns
  Interventions: Behavioral: Session 5
- Session 6 (Experimental): Internalize compassion
  Interventions: Behavioral: Session 6
- Session 7 (Experimental): Me and others - Widening the circle
  Interventions: Behavioral: Session 7
- Session 8 (Experimental): Growing happiness
  Interventions: Behavioral: Session 8
- Session 9 (Experimental): Weaving Wisdom and Compassion into Daily Life
  Interventions: Behavioral: Session 9
- Session 10 (Experimental): Living with Heart
  Interventions: Behavioral: Session 10

INTERVENTIONS:
Behavioral: Session 1 — * Ensuring group interaction, allowing parents to meet each other,
  * Providing information in line with the "Awareness-Based Self-Compassion Training Booklet for Parents of Children with Autism Spectrum Disorder" prepared as training material,
  Arms: Session 1
Behavioral: Session 2 — * Making explanations about the contents of the training sessions to be held with parents,
  * Teaching proper breathing techniques,
  * Visual demonstration and application of relaxation techniques
  Arms: Session 2
Behavioral: Session 3 — * "Breathing break with kindness" application,
  * Thinking and evaluating how threat, impulse and soothing systems develop in individuals' own lives,
  * "Safe place" application,
  * Applying "kindness meditation",
  Arms: Session 3
Behavioral: Session 4 — * "Breathing break with kindness" application,
  * The practice of "establishing a compassionate relationship with resistance",
  * "Kindness meditation: a do-gooder" application,
  * "A hand on the heart" application,
  * "A compassionate companion" application,
  Arms: Session 4
Behavioral: Session 5 — * "Breathing break with kindness" application,
  * The practice of "establishing a compassionate relationship with desire",
  * "Guided meditation to discover the inner pattern" practice,
  * "Kindness meditation: a good friend" application,
  Arms: Session 5
Behavioral: Session 6 — * "Pretending" practice regarding parents' awareness,
  * An expanded version of the practices carried out in previous sessions to raise awareness, the "internalizing compassion" practice,
  * "Kindness meditation: a neutral person", "kindness towards your body" and "walking with kindness" practices, which are based on mindfulness practices and increase body awareness and mindful movement,
  Arms: Session 6
Behavioral: Session 7 — * A "compassionate letter" application, which is carried out by asking parents to think about a situation they have encountered recently or some time ago that still causes distress,
  * "Kindness meditation: the 'difficult' person", "compassion and breathing: yourself" and "compassionate breathing: others" practices,
  * Researching how parents can cope with difficulties and implementing a "compassionate breath break" without words,
  Arms: Session 7
Behavioral: Session 8 — * "Revisiting the good" application to enable parents to experience the five senses in a pleasant way,
  * Practices of "self-forgiveness", "asking for forgiveness", "forgiving others", "gratitude", which can be a way of mending the cracks in parents' relationships with themselves and others,
  * Expanding the practice into "kindness meditation: groups and all beings",
  Arms: Session 8
Behavioral: Session 9 — * The practice of allowing parents to choose a day in their lives for a few minutes to pause mindfully,
  * "A breather for wise and compassionate action" practice,
  * "Calmness meditation" application,
  * "Sharing the joy meditation" application,
  Arms: Session 9
Behavioral: Session 10 — * Evaluating the entire education by telling parents about the practices they can use where help is needed to develop compassion towards self-healing skills,
  * "River of Life" application, which evaluates awareness in depth,
  * Saying goodbye.
  Arms: Session 10

SUMMARY:
Autistic Spectrum Disorder (ASD) is an important public health problem in our country as well as all over the world. The physical, psychological, social and economic problems and mood disorders experienced by the parents of these children can negatively affect not only themselves, but also the effectiveness of the intervention and treatment programs applied to the children. Therefore, many mindfulness-based intervention programs aim to improve stress reduction, resilience and well-being in parents.

In this study, it is aimed to evaluate the effect of mindfulness-based self-compassion training given to parents of children with ASD on stress, resilience and well-being. The research will be carried out with the parents of children aged 7-12 years who applied to the Child and Adolescent Psychiatry Outpatient Clinic of Atatürk University Health Research and Application Center located in Erzurum city center between December 2022 and October 2024 and diagnosed with ASD. The sample of the study was determined by G-power analysis. With the power analysis, it was calculated that at least 68 parents should be included in the sample, in the calculation made at the level of α=0.05, the effect size of 150, 153 (d=0.8) and the power of the study to be 90%. Therefore, the sample size of this study is planned to be 68.

In the collection of research data, an introductory information form containing the socio-demographic data of the child with ASD and the parent, prepared by the researcher in line with the literature, Parental Stress Scale (SIDS), Psychological Resilience Scale for Adults, Warwick-Edinburgh Mental Well-Being Scale, Self-Compassion Scale Short Form (SSS-F), Conscious Awareness Scale (CIFI) will be used.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a developmental disability that can cause a wide variety of difficulties in social interaction, communication, and behavior. ASD is defined in the 5th Edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) as the presence of limited and repetitive behaviors, interests, or activity patterns with the emergence of permanent impairments in social interaction (American Psychiatric Association, 2013). Autism spectrum disorder (ASD) is a lifelong pervasive neurodevelopmental disorder reported to occur in 1 (approximately 2.3%) of 44 8-year-old children in the United States (Alyami et al., 2022; CDC, 2022; Vasilopoulou). and Nisbet, 2016).

Symptoms of ASD vary greatly depending on the child's developmental level and chronological age, and may include a number of behavioral symptoms such as hyperactivity, impulsivity, aggression, self-harming behavior, tantrums, and delayed toilet training (Neff & Faso, 2015; Duarte et al. ., 2005). Supporting children with ASD is often complex, requiring multidisciplinary teamwork and continuity of care (Kohane et al. 2012; Lee et al. 2015). Parents of children with ASD must manage many aspects of caregiving that can be challenging and overwhelming (Bekhet et al., 2012). It has been reported that parents of autistic children experience lower quality of life, more depression, and more pessimism about the future than parents of children with normal development and parents of children with other developmental disabilities (Cappe et al., 2011; Johnson et al., 2011). The number of published studies on the impact of ASD on parents has increased over the past two decades. In a meta-analysis study, it was found that parents of autistic children have higher levels of parenting stress than parents of normally developing children or parents of children with other disabilities (for example, Down syndrome, cerebral palsy, intellectual disability) (Hayes & Watson, 2008). 2013). Severe behavioral symptoms in a child with ASD have been associated with parenting stress, increased depression and anxiety symptoms (Cachia et al., 2016; Junior et al., 2016), and general psychological distress (Keenan et al., 2016). Stigma in social interaction affects well-being and stress in parents caring for a child with ASD (Chan & Lam, 2017; Kinnear et al., 2016; Mak & Kwok, 2010). In addition, it was stated that the well-being of parents was positively affected by social support (Werner & Shulman, 2013).

The severity of a child's autism symptoms and behaviors has consistently been found to be one of the strongest predictors of parental stress (Davis & Carter, 2008; Ingersoll & Hambrick, 2011; Lyons et al., 2010; Hall & Graff, 2012). Children with ASD usually develop anger, aggression, self-harm, tantrums, and repetitive behaviors that are described by parents as destructive, unpredictable, and difficult to manage (Ludlow et al. 2011). Since parents cannot "control" their children due to these situations, they are thought to be misbehaving by strangers and may receive condemnation and disapproval. Parents experience shame due to this situation (Mak & Kwok, 2010; Neff & Faso, 2015).

In a study, it was determined that parenting stress levels should be considered when designing early education interventions for children with ASD. Helping parents of children with ASD reduce their stress levels enables the child to achieve greater gains in time-intensive early education intervention programs (Osborne et al., 2008). Unless parents successfully cope with important stressors and effectively manage mental health problems, the expected effect of behavioral therapies for their children may be low (Osborne et al., 2008), and behavioral problems may increase in children due to parental stress (Lecavalier et al. et al., 2006 ; McGrath, 2013 ; Neece et al., 2012). Self-compassion, which includes being kind to oneself in difficult times, recognizing the common nature of human suffering, and being consciously aware of negative thoughts and emotions, is cited as one of the factors that can be an important coping strategy. Self-compassion includes being open and sensitive to one's emotions in the face of one's own negative experiences, a willingness to reduce the pain arising from these experiences, and approaching oneself with compassion. Self-compassion has three different components: self-compassion, shared experience of humanity, and conscious awareness (Neff, 2003). The "self-compassion" dimension of self-compassion shows the potential of a person to approach one's negative feelings, thoughts, actions or impulses in a forgiving, empathetic, sensitive and patient manner (Gilbert & Irons, 2005).The "common experience of humanity" dimension of self-compassion requires knowing that being human brings with it limited power and that everyone can have flaws and deficiencies. The third dimension of self-compassion, "conscious awareness", includes being able to pay attention to the very moment one is in, clearly and consciously, being aware of and accepting whatever is happening at that moment. Besides being mindful, it is also very important to be able to pay attention to the present moment with compassionate and friendly attention. Mindfulness includes the ability to name and observe the emotions and thoughts one has at the moment, rather than reacting impulsively. In order for an individual to show self-compassion, he must first be aware of his pain (Neff & Tirch, 2013). Awareness requires acknowledging the reality of experiences rather than escaping painful feelings. Therefore, mindfulness is an inevitable component of self-compassion and helps with emotion regulation. Emotion regulation; Being aware of the emotion, intensity and duration of feeling the emotion in the face of negative life experiences (Thompson, 1994). In other words, conscious awareness; It is to be able to provide balanced control of emotions without allowing the individual to accept his painful feelings, but without allowing these feelings to create anxiety in him (Neff, 2003).

In a study conducted with parents of children with ASD, it has been shown that parental stress and well-being are affected by self-compassion (Neff & Faso, 2015; Wong et al., 2016). In a recent study on Mindfulness-Based Stress Reduction (MBSR) and Self-Compassion (SC) training for parents of children with ASD, it was reported that the education applied in parents reduced stress and anxiety and increased their awareness of attention (Rojas-Torres, 2021).

In the literature, international studies on Awareness-Based Self-Compassion training on stress reduction in parents of children with ASD are limited (Rojas-Torres, 2021). International studies on increasing resilience and well-being of Mindfulness-Based Self-Compassion training have not been found. When national surveys were examined, no study was found on the use of Mindfulness-Based Self-Compassion training to reduce stress, increase resilience and well-being. Considering the stress situations experienced by the parents of children with ASD, it is thought that the practice of Awareness-Based Self-Compassion training, as an evidence-based practice, is important for parents regarding stress, resilience and well-being.

ELIGIBILITY:
Inclusion Criteria:

* To be at least a primary school graduate.
* Being the parent of a child whose age is 7-12 and diagnosed with ASD.
* Willingness to participate in the study.
* To be open to communication and cooperation.

Exclusion Criteria:

* Parental psychiatric problems.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | up to 24 hours
  The form consists of 15 questions containing information about the child and his/her parents, created by the researcher within the scope of the literature. The created form includes questions about mother's age, father's age, child's age, age at which the child was diagnosed with ASD, child's gender, child's education level, number of siblings of the child, mother's education level, father's educational status, information about the parents' relationship, and the parent's mental state.
Parental Stress Scale (PASS) | up to 24 hours
  It was developed by Özmen and Özmen (2012) to measure the stress experienced by mothers and fathers in their relationships with their children in daily life. ABSQ consists of a single factor structure consisting of 16 items. The Cronbach alpha coefficient of the scale is .85. The scale is a four-point Likert type (Always=4, Often=3, Sometimes=2, Never=1). The lowest score that can be obtained from the scale is 16, and the highest score is 64. A high score from the scale indicates that parental stress is high.
Resilience Scale for Adults | up to 24 hours
  The dimensions in the scale are called 'self-perception', 'perception of the future', 'structural style', 'social competence', 'family cohesion' and 'social resources'. In the scale, which includes a total of 33 items, a format is used in which positive and negative features are on different sides, and five separate boxes are used for answers in order to avoid biased evaluations in choosing the items. In the schematic evaluation, the scoring method was released in the high or low measurement of psychological resilience.Cronbach Alpha values calculated for the reliability of the scale; It was calculated as 0.76 for 'Self Perception', 0.75 for 'Future Perception', 0.84 for 'Social Competence', 0.89 for 'Family Cohesion', 0.80 for 'Social Resources' and 0.76 for 'Structural Style.
Warwick-Edinburgh Mental Well-Being Scale | up to 24 hours
  Tennant et al. (2007) and adapted into Turkish by Keldal (2015). Consisting of 14 items and a single dimension, this scale covers psychological well-being and subjective well-being and deals with the positive mental health of individuals. The scale is a 5-point Likert type, with a scoring of 1 = strongly disagree, 2 = disagree, 3 = somewhat agree, 4 = agree, 5 = completely agree. A minimum of 14 and a maximum of 70 points are obtained from the scale. High scores obtained from the scale indicate high mental (psychological) well-being. All items of the scale are positive. Cronbach's Alpha internal consistency reliability coefficient was found to be 0.92.
Self-Compassion Scale Short Form (STS-C) | up to 24 hours
  The scale developed by Neff (2003) was validated and reliable in Turkish by Yıldırım and Sarı in 2018. The scale was confirmed to have a structure consisting of 11 items, a single dimension and two complementary components (positive component and negative component). The internal consistency coefficient of the scale was calculated as .75. Neff (2014) used the scale he developed in parents with children with ASD and reported that self-compassion can play an important role in the well-being of parents of children with autism. SSS-F It is recommended to be used in studies where total score will be used to measure self-compassion.
Conscious Awareness Scale (CIFS) | up to 24 hours
  It was developed by Brown and Ryan (2003) in order to evaluate the CP level of individuals. In the study of Ozgreen et al. (2011), its Turkish validity and reliability were performed. The scale is a one-dimensional, six-point Likert-type scale consisting of 15 questions. The Cronbach's alpha coefficient of the scale was found to be 0.80. The minimum and maximum points that individuals can get from the scale are between 15 and 90. High scores indicate a high BF level.

CONTACTS AND LOCATIONS:
Overall Officials: DİLEK KILIÇ, Study Director — Atatürk University, Faculty of Nursing
Locations (1):
- Ataturk University Faculty of Nursing, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No